CLINICAL TRIAL: NCT06802276
Title: Employing Smart Underwear to Measure Gut Microbial Hydrogen Sulfide Production
Brief Title: Smart Underwear to Measure Diet-Induced Hydrogen Sulfide Production
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); University of Maryland, College Park (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 24-1861; R33DK132310-03 (NIH)
Record Dates: First submitted 2025-01-15; First posted 2025-01-31 (Actual); Last update posted 2025-05-26 (Actual); Status verified 2025-03

CONDITIONS: Hydrogen Sulfide; Gastrointestinal Microbiome
Keywords: Hydrogen Sulfide; H2S; Diet; Cysteine; Gut Microbiome

STUDY DESIGN:
Intervention Model Description: The study design is a two-period crossover feeding study, in which participants will be randomly assigned to each of a high cysteine and low cysteine isocaloric diet for a 6-day period each. Additionally, a 3-day baseline period will occur prior to each dietary intervention period. Diet intervention periods will be separated by a washout period. This washout period may vary slightly between participants and will last for a minimum of 9 days and a maximum of 13 days.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigators and the outcomes assessors will not know which order of diets the participant has been assigned. The participant will not be explicitly told which diet he or she is receiving during each period, but by the nature of the differences between the high cystine and low cystine diets, the participant may be able to guess based on the menus.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Cysteine Diet (Active Comparator): A dietary pattern designed to have a high level of dietary cysteine
  Interventions: Other: High Cysteine Diet
- Low Cysteine Diet (Other): A dietary pattern designed to have a low level of dietary cysteine
  Interventions: Other: Low Cysteine Diet

INTERVENTIONS:
Other: High Cysteine Diet — A healthy diet pattern which contains high levels of cysteine or cysteine-related compounds. The high and low cysteine diets will be designed by a research dietician to differ primarily in their concentration of cysteine while providing similar levels of calories, protein, fats, carbohydrates, fiber, and several micronutrients. No additional supplementation of cysteine will be used. Examples of high cysteine foods: chicken, eggs, lentils, yogurt, garlic, cheese, soybeans
  Arms: High Cysteine Diet
Other: Low Cysteine Diet — A healthy diet pattern which contains low levels of cysteine or cysteine-related compounds. The high and low cysteine diets will be designed by a research dietician to differ primarily in their concentration of cysteine while providing similar levels of calories, protein, fats, carbohydrates, fiber, and several micronutrients. The low cysteine diet includes lower-protein food sources. Examples of low cysteine foods: rice, bread, oranges, bananas, lettuce, snow peas, peppers
  Arms: Low Cysteine Diet

SUMMARY:
The purpose of this study is to evaluate the ability of a wearable Smart Underwear prototype device to quantify diet-induced changes in gut microbial hydrogen sulfide (H₂S) production. The core design is a single-site, 2-period, crossover feeding study with 6-day diet periods and an approximately 11-day washout period. Participants are fed each of two isocaloric diets designed to contrast gut microbial H₂S production (i.e., a high cysteine vs. low cysteine diet), in a random order.

DETAILED DESCRIPTION:
H₂S is a circulating signaling molecule that plays numerous roles in human physiology. H₂S produced exogenously by the gut microbiota influences human health by modulating systemic H₂S bioavailability in a diet-dependent manner. Several lines of evidence suggest excessive gut microbial H₂S production may be etiologically involved in a wide range of diseases, from colorectal cancer to ulcerative colitis. However, research on the health-relevant effects of gut microbially-produced H₂S has been constrained by technical limitations.

Gap: Current techniques for measuring gut microbial H₂S production are imprecise, invasive, and have limited temporal resolution, hindering the ability to deconvolute how gut microbial H₂S production both affects human health and is influenced by factors such as diet. Gaseous rectal effluent (flatus) is an ideal, yet untapped biospecimen to measure gut microbial H₂S production.

Preliminary Evidence: To enable real time measurements of gut microbial H₂S production in flatus, the investigators are developing a wearable device called "Smart Underwear". The Smart Underwear device is fundamentally different from previous methods used to measure gut microbial H₂S production. The Smart Underwear device uses an array of metal oxide gas sensors coupled with a multi-layer filtration system to selectively measure H₂S by comparing the signal from filtered and unfiltered sensors. The Smart Underwear sensor array is adhered to the outside of a participant's underwear adjacent to the perineum. Through in vitro and human wearing validation, the investigators have demonstrated the feasibility of the Smart Underwear v1 prototype to measure gut microbial H₂S production in flatus and have shown that the device has potential utility in human cohort studies as a non-invasive device.

The long-term goal of this study is to develop a validated Smart Underwear device that measures real time gut microbial hydrogen sulfide (H₂S) production which is responsive to dietary changes and capable of predicting of pathophysiological outcomes.

The investigators will validate the Smart Underwear prototype device using structured dietary modulation of H₂S production.

Aim: Conduct a randomized controlled feeding trial to evaluate the ability of the Smart Underwear device to quantify diet-induced changes in gut microbial H₂S production.

Hypothesis: The investigators hypothesize that the Smart Underwear device will detect higher H₂S concentrations in flatus during a high cysteine dietary intervention compared to a low cysteine dietary intervention.

Methods: The investigators will employ a randomized crossover feeding trial with two arms designed to contrast gut microbial H₂S production by modulating dietary cysteine while controlling other dietary factors (total calories and nutrients). The investigators have conducted extensive background research to determine that modulation of dietary cysteine is the most effective means of producing a diet-induced contrast in H₂S production. Participants will wear the Smart Underwear device during the dietary interventions allowing for a rigorous evaluation of the devices ability to detect diet-induced alterations of gut microbial H₂S production in flatus.

ELIGIBILITY:
The inclusion/exclusion criteria will identify generally healthy volunteers that are able to ingest the intervention diets. Exclusion criteria based on diseases, medications, allergies, and specific dietary requirements will minimize the risks of adverse reactions to the intervention diets.

Inclusion Criteria:

* Generally healthy volunteers defined as having no major known health conditions (e.g., diabetes, cancer, hypertension, etc.).
* Normal bowel movements, with approximately 1 bowel movement reported per day
* Willing to discuss flatus
* Ages >18yrs
* Willing to complete the entire study protocol, i.e. eating all of the food that is provided and completing all required measurements.

Exclusion Criteria:

* Self-report or other evidence of diabetes, other endocrine/metabolic abnormality, dyslipidemia, morbid obesity, severe hypertension, chronic kidney disease, liver disease, pulmonary disease, gastrointestinal, and cardiovascular diseases
* Chronic medications for any of the above conditions
* Food allergy that interferes with ability to complete the study
* Food preferences, intolerance, or dietary requirements that would interfere with diet adherence
* Planned dietary changes during the study period
* Lack of appropriate food refrigeration and preparation equipment (e.g.- oven or microwave)
* Pregnancy or planned pregnancy in the next month
* Physical measurements: BMI > 35 kg/m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-05-21 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Hydrogen sulfide (H2S) | Daily for 6 days during each dietary intervention period (total of 12 days).
  Participants will be instructed to wear the Smart Underwear device for all waking hours during the baseline and feeding periods except for bathing and exercise. The Smart Underwear device does not need to be worn while sleeping due to the decreased frequency of flatus. Participants will be warned by the Smart Underwear device if the device is not worn for at least 12 hours per day or if the device detects that it is being worn incorrectly. Aggregate metrics from the device will be included in either the on-site or virtual discussions with staff.

SECONDARY OUTCOMES:
Microbiome Activity Index | Daily for 6 days during each dietary intervention period (total of 12 days).
  A high gut microbiome activity is closely correlated with hydrogen gas production, reflected in the increase of both flatus frequency and hydrogen concentration (e.g., accumulated gas can be expelled in a few high-intensity events or through a series of smaller flatus). The investigators derived a Microbiome Activity Index which combines information on the rate of change in hydrogen and hydrogen sulfide, number of flatus events, and time between flatus events.
Gastrointestinal Microbiome | The final day of each 6-day dietary intervention period (total of 2 days).
  Participants will self-collect fecal samples using the OMNIgut OM-200 and OM-205 kits.100 Microbiome Sample Collection Kits. Shotgun metagenomic sequencing will be performed to measure changes in microbiome composition and diversity.
Experienced Symptoms Questionnaire | The final day of each 6-day dietary intervention period (total of 2 days).
  Participants will complete a questionnaire about symptoms experienced while on each diet, including symptoms related to fall risk (e.g., feeling faint), food intake and output (e.g., bloating, constipation), fluid intake and output (e.g., excessive thirst), and general symptoms (e.g., fatigue or low energy). Participants will be asked to rate each listed symptom as: did not occur, mild, moderate, or severe. Score range 0-67, higher score worse symptoms.
Participant Wearing Time | Daily for 6 days during each dietary intervention period (total of 12 days).
  How long participants wear the Smart Underwear device. Participants will be instructed to wear the Smart Underwear device for all waking hours during the feeding intervention periods except during bathing and exercise. The Smart Underwear device does not need to be worn while sleeping due to the decreased frequency of flatus. The Smart Underwear device internally detects and records wear time; aggregated wear time metrics will be collected from the device at the end of each intervention period.
Systolic Blood Pressure (SBP) | The final day of each 6-day dietary intervention period (total of 2 days).
  Following 5 minutes of resting in a seated position, blood pressure will be measured in triplicate, and the average of the last two readings (in mmHg) will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Noel T Mueller, PhD, Principal Investigator — University of Colorado, Denver; Andrew B Hall, PhD, Principal Investigator — University of Maryland, College Park
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States